CLINICAL TRIAL: NCT03400917
Title: Phase II Trial of Autologous Dendritic Cells Loaded With Autologous Tumor Associated Antigens (AV-GBM-1) as an Adjunctive Therapy Following Primary Surgery Plus Concurrent Chemoradiation in Patients With Newly Diagnosed Glioblastoma
Brief Title: Autologous Dendritic Cells Loaded With Autologous Tumor Associated Antigens for Treatment of Newly Diagnosed Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aivita Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-GBM-P01
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Newly Diagnosed Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AV-GBM-1 (Experimental): Autologous dendritic cells loaded with tumor associated antigens from a short-term cell culture of autologous tumor cells. AV-GBM-1 is admixed with granulocyte-macrophage colony stimulating factor (GM-CSF) as an adjuvant, prior to injection.
  Interventions: Biological: AV-GBM-1

INTERVENTIONS:
Biological: AV-GBM-1 — Investigational treatment with AV-GBM-1

SUMMARY:
This is a single-arm, open-label phase II clinical trial in which approximately 55 patients with newly diagnosed glioblastoma (GBM) will be enrolled with the intent to receive an autologous dendritic cell vaccine consisting of autologous dendritic cells loaded with autologous tumor-associated antigens (AV-GBM-1).

DETAILED DESCRIPTION:
This is a single-arm, open-label phase II clinical trial in which approximately 55 patients will be enrolled with the intent to receive AV-GBM-1. Patients eligible for treatment will be those (1) who have recovered from surgery such that they are about to begin concurrent chemotherapy and radiation therapy (CT/RT), (2) for whom an autologous tumor cell line has been established, (3) have a KPS of > 70, and (4) have undergone successful leukapheresis from which peripheral blood mononuclear cells (PBMC) were obtained that can be used to generate dendritic cells (DC).

The primary endpoint of this trial is overall survival (OS), death from any cause measured from the date of study enrollment for treatment with AV-GBM-1. Secondary endpoints will include (1) PFS measured from date of enrollment, (2) OS/PFS measured from date of diagnosis and (3) OS/PFS from date of enrollment based on KPS, age, and extent of surgical resection. Tertiary endpoints will include (1) OS/PFS from date of first injection and (2) OS/PFS from date of first injection in patients who completed concurrent CT/RT and had not progressed.

Patient Population: Patients 18 years or older with newly diagnosed glioblastoma [World Health Organization (WHO) Grade IV glioma, Grade IV anaplastic astrocytoma, glioblastoma or gliosarcoma, glioblastoma multiforme (GBM)] who have recovered from surgery, for whom an autologous tumor cell culture and leukapheresis product are available, who have a KPS of > 70, and who are about to begin concurrent CT/RT.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Score of 70-100%
* Histology confirmed to be GBM (Grade IV WHO, glioblastoma, gliosarcoma)
* Successful establishment of an autologous cancer cell line by AIVITA Biomedical, Inc.
* Collection of a satisfactory leukapheresis product
* About to begin concurrent CT/RT
* Given written informed consent to participate in the study

Exclusion Criteria:

* Known to have active hepatitis B or C or HIV
* Karnofsky Performance Score of < 70%
* Known underlying cardiac disease associated with myocardial dysfunction that requires active medical treatment, or unstable angina related to atherosclerotic cardiovascular disease, or under treatment for arterial or venous peripheral vascular disease
* Diagnosis of any other invasive cancer or other disease process which is considered to be life-threatening within the next five years, and/or taking anti-cancer therapy for cancer other than GBM
* Active infection or other active medical condition that could be eminently life-threatening, including active blood clotting or bleeding diathesis.
* Known autoimmune disease, immunodeficiency, or disease process that involves the chronic use of immunosuppressive therapy.
* Received another investigational drug within 28 days of the first dose or are planning to receive another investigational drug while receiving this investigational treatment.
* Known hypersensitivity to GM-CSF
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Overall Survival | 3 years
  Overall Survival: time to death from date of enrollment for intent-to-treat with AV-GBM-1

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Dillman, MD, Study Chair — Aivita Biomedical, Inc.
Locations (8):
- United States (8):
  - Scripps Health, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UC Irvine Medical Center, Orange, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Norton Cancer Institute, Louisville, Kentucky
  - Rutgers Cancer Institute, New Brunswick, New Jersey

REFERENCES:
- [Derived] Bota DA, Taylor TH, Piccioni DE, Duma CM, LaRocca RV, Kesari S, Carrillo JA, Abedi M, Aiken RD, Hsu FPK, Kong XT, Hsieh C, Bota PG, Nistor GI, Keirstead HS, Dillman RO. Phase 2 study of AV-GBM-1 (a tumor-initiating cell targeted dendritic cell vaccine) in newly diagnosed Glioblastoma patients: safety and efficacy assessment. J Exp Clin Cancer Res. 2022 Dec 14;41(1):344. doi: 10.1186/s13046-022-02552-6. PMID 36517865